CLINICAL TRIAL: NCT00396773
Title: Neonatal Brain Waves After Electrocoagulation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: Elactrobrainwaves-HMO-CTIL
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2006-11-10 (Estimated); Status verified 2006-11

CONDITIONS: Epilepsy
Keywords: electrocoagulation,pregnancy,brian waves
MeSH Terms: conditions — Epilepsy; Hyperthermia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Electrocoagulation effect of neonatal brain waves after cesarean section

DETAILED DESCRIPTION:
Electrocoagulation is used for bleeding control on usual basis in cesarean sections and other surgical procedures .

We are planning to test the effect of electrocoagulation unipolar on neonatal brain waves compared with neonates that were exposed to bipolar electrocoagulation .Bipolar electrocoagulation should have les of an effect because of it coagulates in a close ,closed electrical cycle .

ELIGIBILITY:
Inclusion Criteria:

* term normal newborn after normal pregnancy after elective cesarean section

Exclusion Criteria:

* any fetal or neonatal disease or condition that may affect brain waves

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Study Completion 2008-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, Principal Investigator — Hadassah University Medical Organization
Locations (1):
- Contact Arik Tzukert,DMD, Jerusalem, Israel

REFERENCES:
- [Background] Rosen I. The physiological basis for continuous electroencephalogram monitoring in the neonate. Clin Perinatol. 2006 Sep;33(3):593-611, v. doi: 10.1016/j.clp.2006.06.013. PMID 16950313